CLINICAL TRIAL: NCT00595985
Title: Phase II Trial of Sorafenib as Second Line Therapy in Patients With Advanced or Metastatic Gastric Cancer
Brief Title: Sorafenib as a Second Line Treatment in Patients With Advanced or Metastatic Gastric Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low response rate, no evidence of PFS or OS improved.
Sponsor: Fudan University (Other)
Responsible Party: Base for drug clinical trials, Fudan University cancer hospital, Department of medical oncology, Cancer Hospital, Fuandan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sorafenib-MGC
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Gastric Cancer
Keywords: Time to Progression; Toxicity; Overall survival; Response rate; Quality of live; Toxicities
MeSH Terms: conditions — Stomach Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): administer sorafenib 400mg bid until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — sorafenib 400mg bid, and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Other Names: treatment group

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of sorafenib as second line treatment in patients with Advanced or Metastatic Gastric Cancer (A/MGC).

DETAILED DESCRIPTION:
Up to now, although FU based, cisplatin based and taxane based regimen, and ECF regimen have been suggested as the first line therapy for A/MGC by FDA, there is no standard regimen for patients with A/MGC as second line treatment. Based on the promising results of sorafenib in primary hepatic carcinoma and renal cancer, we design this clinical trial to evaluate the efficacy, time to progression and overall survival of sorafenib for A/MGC patients as a second line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic adenocarcinoma of the stomach
* ECOG performance scale ≤ 2
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan)
* Adequate hepatic, renal, heart, and hematologic functions:

  * platelets>80 × 109/L
  * neutrophil>2.0 × 109/L
  * serum creatinine ≤ 1.5mg/dl
  * total bilirubin within upper limit of normal(ULN)
  * serum transaminase ≤ 2.5 × the ULN

Exclusion Criteria:

* Pregnant or lactating women
* Concurrent cancer
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Neuropathy, brain, or leptomeningeal involvement
* Uncontrolled significant comorbid conditions and previous radiotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
time to progression | every six weeks

SECONDARY OUTCOMES:
toxicity | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China